CLINICAL TRIAL: NCT03066492
Title: Evaluation of a Novel Hospital Discharge Clinic to Improve Care Coordination and Reduce Rehospitalization Among Low Income Adults
Brief Title: Evaluation of a Hospital Discharge Clinic to Improve Care Coordination and Reduce Rehospitalization in Low Income Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ronald Ackermann, Senior Associate Dean for Public Health, Director, Institute for Public Health and Medicine, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00200259
Record Dates: First submitted 2017-02-22; First posted 2017-02-28 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Patient Readmission
Keywords: Tertiary Care Center; Patient Readmission; Health Services Research; Hospital Readmissions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Federally Qualified Health Center (Active Comparator): Each patient is provided with information by telephone and mail, offering assistance to receive a follow-up appointment at a nearby Federally Qualified Health Center.
  Interventions: Other: Federally Qualified Health Center
- Northwestern Follow Up Care Coordination (Experimental): Each patient is provided with information by telephone and mail, offering assistance to receive a follow-up appointment at the Northwestern Transitional Care Follow Up Clinic.
  Interventions: Other: Northwestern Follow Up Care Coordination

INTERVENTIONS:
Other: Northwestern Follow Up Care Coordination — Each patient is provided with information by telephone and mail, offering assistance to receive a follow-up appointment at the Northwestern Transitional Care Follow Up Clinic.
  Arms: Northwestern Follow Up Care Coordination
Other: Federally Qualified Health Center — Each patient is provided with information by telephone and mail, offering assistance to receive a follow-up appointment at a nearby Federally Qualified Health Center.
  Arms: Federally Qualified Health Center

SUMMARY:
This randomized controlled trial examines the effects of a transitional care clinic for high-risk patients at an academic medical center who had no trusted medical home. The trial will provide the first reliable evaluation of the Northwestern Transitional Care Clinic / Follow Up Clinic's (NFC) impact on re-admissions, care coordination, and costs. This research will allow us to assess the value of the NFC and similar models of care for providing a more coordinated care approach that results in better treatment outcomes for urban poor populations.

It is hypothesized that NFC patients will have fewer 90-day re-hospitalizations and are more likely to have a usual source of primary care 6 months after discharge.

DETAILED DESCRIPTION:
The Northwestern Transitional Care Follow-up Clinic (NFC) was established in 2012 to improve the coordination of care for these patients following inpatient or Emergency Department discharge from Northwestern Memorial Hospital. Since 2012, the NFC has constructed an integrated team care approach, logging about 2000 post-discharge encounters with Medicaid or patients without insurance. The NFC model has evolved over the past 2 years in response to a need to address mental as well as physical health needs and to interface with community resources to address social determinants of health that might otherwise lead to frequent re-admission. By working with clinical partners and public payers like Medicaid and County Care, the NFC has also worked to transition patients to accessible primary care medical homes that will provide behavioral, physical, and preventive care. The current study will provide the first reliable evaluation of the clinic's impact on re-admissions, care coordination, and costs. This research will allow us to assess the value of the NFC and similar models of care for providing a more coordinated care approach that results in better treatment outcomes for urban poor populations.

ELIGIBILITY:
Inclusion Criteria:

* All patients eligible for Northwestern Transitional Follow Up care post-discharge from Northwestern Memorial Hospital
* Adults (18 years of age or older)
* Patients referred by an Northwestern Memorial Hospital care provider for discharge coordination by the Northwestern Transitional Follow Up Clinic

Exclusion Criteria:

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant Women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
90-Day Re-hospitalization or Death | 90 days
  90-day re-hospitalization (Emergency Department and/or inpatient admission) or death

SECONDARY OUTCOMES:
Usual Source of Primary Care | 6 months
  Patient report of being seen in a usual source of primary medical care 6 months after discharge
30-Day Re-hospitalization or Death | 30 days
  90-day re-hospitalization (Emergency Department and/or inpatient admission) or death
180-Day Re-hospitalization or Death | 180 days
  180-day re-hospitalization (Emergency Department and/or inpatient admission) or death
365-Day Re-hospitalization or Death | 365 days
  365-day re-hospitalization (Emergency Department and/or inpatient admission) or death
Health Advocate Effect | 12 months
  This evaluation will determine if being offered support of a novel care team member known as a "health advocate" (a form of care navigator who will assist patients to overcome social determinants of readmission) is more likely to prevent hospital readmission than receiving the standard Northwestern Transitional Follow Up Care team intervention alone.
Intervention Cost | 12 months
  This is an evaluation of the incremental costs to implement and sustain standard Northwestern Transitional Follow Up team care, as well as the enhanced standard + health advocate personnel model

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Ackermann, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liss DT, Ackermann RT, Cooper A, Finch EA, Hurt C, Lancki N, Rogers A, Sheth A, Teter C, Schaeffer C. Effects of a Transitional Care Practice for a Vulnerable Population: a Pragmatic, Randomized Comparative Effectiveness Trial. J Gen Intern Med. 2019 Sep;34(9):1758-1765. doi: 10.1007/s11606-019-05078-4. Epub 2019 May 29. PMID 31144279
- [Derived] Ackermann RT, Liss DT, French DD, Cooper AJ, Aikman C, Schaeffer C. Randomized Trial Evaluating Health System Expenditures with Transitional Care Services for Adults with No Usual Source of Care at Discharge. J Gen Intern Med. 2022 Nov;37(15):3832-3838. doi: 10.1007/s11606-022-07473-w. Epub 2022 Mar 9. PMID 35266127